CLINICAL TRIAL: NCT00054119
Title: A Phase II Evaluation of Karenitecin in the Third-Line Treatment of Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Karenitecin in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0186D; NCI-2012-02514 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000269898; BIONUM-KTN22307; GOG-0186D (Other: Gynecologic Oncology Group); GOG-0186D (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Primary Peritoneal Carcinoma; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — cositecan

ARMS (1):
- Treatment (Experimental): Patients receive karenitecin IV over 1 hour on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cositecan; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cositecan — Given IV
  Other Names: BNP1350; DB 172; Karenitecin
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of karenitecin in treating patients who have persistent or recurrent ovarian epithelial cancer or primary peritoneal cancer that has not responded to platinum-based treatment. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the antitumor activity of karenitecin in patients with persistent or recurrent platinum-resistant ovarian epithelial or primary peritoneal cancer.

II. Determine the toxicity of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive karenitecin IV over 1 hour on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial or primary peritoneal cancer

  * Recurrent or persistent disease
  * Platinum-resistant disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* At least 1 target lesion to assess response (tumors within a previously irradiated field are designated as non-target)
* Ineligible for a higher priority GOG study or other phase II cytotoxic study for platinum-resistant disease
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No myocardial infarction within the past 6 months
* No cerebrovascular accident within the past 6 months
* No transient ischemic attack within the past 6 months
* No uncontrolled hypertension
* No decompensated or uncontrolled chronic heart failure
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No neuropathy (sensory or motor) grade 2 or greater
* No other invasive malignancies within the past 5 years except nonmelanoma skin cancer
* No active infection requiring antibiotics
* At least 3 weeks since prior biological or immunological agents
* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered
* No more than 2 prior cytotoxic chemotherapy regimens, with no more than 1 non-platinum, non-taxane regimen
* No prior karenitecin or camptothecin analogue/derivative
* At least 1 week since prior hormonal therapy

  * Concurrent hormone replacement therapy allowed
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 25% of marrow-bearing areas
* Recovered from recent surgery
* At least 3 weeks since prior therapy directed at this malignancy
* No prior anticancer therapy that would preclude study therapy
* No concurrent amifostine or other protective reagents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-01; Primary Completion 2005-09-30 (Actual)

PRIMARY OUTCOMES:
Frequency of objective response | Up to 6 years
Duration of objective response | Up to 6 years
Frequency of observed adverse effects, graded according to CTC version 2.0 | Up to 6 years
Severity of observed adverse effects, graded according to CTC version 2.0 | Up to 6 years
Survival time for all patients | Up to 6 years
Duration of progression-free interval for all patients | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: John Kavanagh, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group of Arizona, Phoenix, Arizona, United States